CLINICAL TRIAL: NCT04161859
Title: Observational Study on the Use of the Nutraceutical With Cardio-metabolic Actions in the Patient in Primary and Secondary Prevention
Brief Title: Use of Nutraceuticals in Clinical Practice
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Principal Investigator, University of Pavia
Other Study IDs: P-20160020534
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Dyslipidemias; Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2; Hypertension | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Nutraceutical — Nutraceutical with action on glycemia, dsylipidemia or hypertension will be considered.

SUMMARY:
The aim of this study will be to evaluate the use of the nutraceutical with cardio-metabolic actions in clinical practice in addition to a Mediterranean diet scheme, normally recommended in the clinic. In particular the study will analyze how much the nutraceutical is prescribed and what are the purposes for which it is used and at what dosages.

DETAILED DESCRIPTION:
The aim of this study will be to evaluate the use of the nutraceutical with cardio-metabolic actions in clinical practice in addition to a Mediterranean diet scheme, normally recommended in the clinic. In particular the study will analyze how much the nutraceutical is prescribed and what are the purposes for which it is used and at what dosages. In particular, attention will be focused on the following substances: berberine (500-1000 mg/day), monacolin (5-10 mg/day), phytosterols (0.9-1.8 g/day), resveratrol (100-500 mg/day), omega-3 (1-3 g/day), alpha lipoic acid (400-800 mg/day), curcumin (400 mg/day), psyllum (3.5 g/day), coenzyme Q10 (100-200 mg/day), inositol (250-600 mg/day), glucomannan (1-4 g/day), chitosan (800-1200 mg/day), guar fiber (10-20 g/day), L-arginine (250 mg/day).

ELIGIBILITY:
Inclusion Criteria:

Diabetic patients in primary and secondary prevention or Hypertensive patients in primary and secondary prevention or Dyslipidemic patients in primary and secondary prevention

Exclusion Criteria:

Patients with hystory of malignancy, and significant neurological or psychiatric disturbances, including alcohol or drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic, or hypertensive or dyslipidemic patients in primary and secondary prevention
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of the use of nutraceutical in clinical practice | From 2010 to 2015
  Prevalence

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy